CLINICAL TRIAL: NCT01538680
Title: An Open-label Phase IIIb Study of Regorafenib in Patients With Metastatic Colorectal Cancer (CRC) Who Have Progressed After Standard Therapy
Brief Title: Regorafenib in Subjects With Metastatic Colorectal Cancer (CRC) Who Have Progressed After Standard Therapy
Acronym: CONSIGN
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15967; 2011-005836-25 (EudraCT Number)
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) — Subjects will receive 160 mg regorafenib po every day (qd) for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off). Subjects will continue on treatment until at least one of the following occurs (main criteria):
  Progressive Disease (PD). The subject may continue treatment at the investigator's discretion.
  Death Unacceptable toxicity Subject withdraws consent Treating physician determines discontinuation of treatment is in the subject's best interest Substantial non-compliance with the protocol

SUMMARY:
This is a phase III B, prospective, interventional, open-label, single-arm, multicenter study to provide regorafenib to subjects diagnosed with metastatic colorectal cancer who have failed after standard therapy and for whom no therapy alternatives exist, in the time between positive results and approval / availability on the market, and to collect safety data for regorafenib until market access.

Regorafenib is an oral (i.e. taken by mouth) multi-targeted kinase inhibitor. A kinase inhibitor targets certain key proteins that are essential for the survival of the cancer cell. By specifically targeting these proteins, regorafenib may stop cancer growth. The growth of the tumor may be decreased by preventing these specific proteins from functioning.

The primary endpoint of this study will be safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age
* Life expectancy of at least 3 months
* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Subjects with metastatic colorectal cancer (Stage IV)
* Progression during or within 3 months following the last administration of approved standard therapies which must include fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab and cetuximab/panitumumab (if KRAS WT) (WT: wild type)
* ECOG Performance Status of ≤ 1 (ECOG: Eastern Cooperative Oncology Group)
* Adequate bone marrow, liver and renal function
* Women of childbearing potential and men must agree to use adequate contraception

Exclusion Criteria:

* Prior treatment with regorafenib
* Congestive heart failure >/= New York Heart Association (NYHA) class 2
* Uncontrolled hypertension (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management)
* Any hemorrhage or bleeding event >/= CTCAE Grade 3 within 4 weeks prior to the start of study medication.
* Persistent proteinuria of CTCAE Grade 3 (>3.5g/24 hours)
* Unresolved toxicity higher than CTCAE (v. 4.0) Grade 1 attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin induced neurotoxicity </= Grade 2
* Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 weeks (or within 6 weeks for mitomycin C) before starting to receive study medication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (182):
- United States (56):
  - Duarte, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Orange, California
  - Santa Maria, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Jacksonville, Florida
  - Miami Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Park Ridge, Illinois
  - Cedar Rapids, Iowa
  - Sioux City, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Brewer, Maine
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - Jefferson City, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Lake Success, New York
  - New York, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Sumter, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Temple, Texas
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Australia (5):
  - Concord, New South Wales
  - St Leonards, New South Wales
  - Woodville South, South Australia
  - Footscray, Victoria
  - Parkville, Victoria
- Austria (4):
  - Graz, Styria
  - Innsbruck, Tyrol
  - Wels, Upper Austria
  - Vienna
- Belgium (4):
  - Bruxelles - Brussel
  - Edegem
  - Leuven
  - Roeselare
- Canada (7):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Mississauga, Ontario
  - Oshawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec
- Czechia (2):
  - Brno
  - Prague
- Denmark (2):
  - Aarhus C
  - Copenhagen
- Finland (2):
  - Helsinki
  - HUS
- France (13):
  - Avignon
  - Bordeaux
  - Clermont-Ferrand
  - Le Mans
  - Lille
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Reims
  - Saint-Herblain
  - Strasbourg
  - Toulouse
- Germany (23):
  - Esslingen am Neckar, Baden-Wurttemberg
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Hanover, Lower Saxony
  - Oldenburg, Lower Saxony
  - Bochum, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Herne, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Porta Westfalica, North Rhine-Westphalia
  - Recklinghausen, North Rhine-Westphalia
  - Trier, Rhineland-Palatinate
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Hamburg
- Greece (2):
  - Heraklion
  - Kifissia / Athens
- Budapest, Hungary
- Ireland (2):
  - Cork
  - Dublin
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (13):
  - Foggia, Apulia
  - Napoli, Campania
  - Modena, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Brescia, Lombardy
  - Milan, Lombardy
  - Palermo, Sicily
  - Ancona, The Marches
  - Florence, Tuscany
  - Pisa, Tuscany
  - Padua, Veneto
- Mexico (8):
  - Irapuato, Guanajuato
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - México, D.F., Mexico City
  - Aguascalientes
  - Oaxaca City
  - Toluca
  - Veracruz
- Netherlands (2):
  - Amsterdam
  - Leiden
- Oslo, Norway
- Poland (2):
  - Bialystok
  - Poznan
- Portugal (2):
  - Coimbra
  - Porto
- Russia (6):
  - Kazan'
  - Krasnodar
  - Moscow
  - Obninsk
  - Orenburg
  - Saint Petersburg
- Spain (11):
  - Córdoba, Andalusia
  - Badalona (Barcelona), Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Sabadell, Barcelona
  - Santander, Cantabria
  - A Coruña
  - Barcelona
  - Madrid
  - Málaga
  - Seville
  - Valencia
- Sweden (2):
  - Linköping
  - Uppsala
- Switzerland (5):
  - Basel, Canton of Basel-City
  - Chur, Kanton Graubünden
  - Bern
  - Geneva
  - Zurich
- United Kingdom (2):
  - Leicester, Leicestershire
  - Manchester

REFERENCES:
- [Derived] Cervantes A, Tabernero J, Garcia-Carbonero R, Sastre J, Feliu J, Carmen Guillen-Ponce, Paredes BG, Carral A, Munoz J. Regorafenib in patients with metastatic colorectal cancer in Spain: from clinical trials to real-world evidence. Future Oncol. 2024;20(20):1401-1413. doi: 10.1080/14796694.2024.2340422. Epub 2024 Jun 11. PMID 38861286
- [Derived] Van Cutsem E, Martinelli E, Cascinu S, Sobrero A, Banzi M, Seitz JF, Barone C, Ychou M, Peeters M, Brenner B, Hofheinz RD, Maiello E, Andre T, Spallanzani A, Garcia-Carbonero R, Arriaga YE, Verma U, Grothey A, Kappeler C, Miriyala A, Kalmus J, Falcone A, Zaniboni A. Regorafenib for Patients with Metastatic Colorectal Cancer Who Progressed After Standard Therapy: Results of the Large, Single-Arm, Open-Label Phase IIIb CONSIGN Study. Oncologist. 2019 Feb;24(2):185-192. doi: 10.1634/theoncologist.2018-0072. Epub 2018 Sep 6. PMID 30190299
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/